CLINICAL TRIAL: NCT06504082
Title: Comparison of the Effectiveness of Single-Dose Methotrexate Protocol With Letrozole + Single-Dose Methotrexate in the Medical Treatment of Patients Diagnosed With Ectopic Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Metin Ayğar, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YuzuncuYıl_MTX_LTZ
Record Dates: First submitted 2024-06-30; First posted 2024-07-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Ectopic Pregnancy
Keywords: methotrexate; letrozole
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Letrozole; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole + Single-Dose Methotrexate Group (Active Comparator): Patients in the MTX + letrozole group received letrozole tablets (Femara 2.5 mg) once daily for ten days starting from the day of MTX administration.
  Interventions: Drug: Letrozole
- Single-Dose Methotrexate (Active Comparator): After confirming the diagnosis of tubal ectopic pregnancy, each patient received a single dose of intramuscular MTX (50 mg/m² MTX) on the same day.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Letrozole — Patients in the MTX + letrozole group received letrozole tablets (Femara 2.5 mg) once daily for ten days starting from the day of MTX administration.
  Arms: Letrozole + Single-Dose Methotrexate Group
Drug: Methotrexate — After confirming the diagnosis of tubal ectopic pregnancy, each patient will receive a single dose of intramuscular MTX (50 mg/m² MTX) on the same day
  Arms: Single-Dose Methotrexate

SUMMARY:
The objective of the study is to compare the effectiveness of single-dose methotrexate and letrozole + single-dose methotrexate in treating ectopic pregnancy, focusing on treatment success, changes in ß-hCG levels, hemogram and biochemical markers, surgical intervention due to rupture, fertility preservation, and reduction of maternal morbidity, mortality, and healthcare costs. This is a prospective study conducted on 60 ectopic pregnancy patients at Van Yuzuncu Yil University from June 2021 to September 2022. Thirty patients received single-dose methotrexate, while the other thirty received letrozole + single-dose methotrexate. Inclusion criteria were ß-hCG <5000 mIU/mL, ectopic mass <3-4 cm, no persistent abdominal pain, no fetal cardiac activity, and no contraindications to the treatments. Outcomes measured included treatment success, blood parameter changes, and the need for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ectopic pregnancy according to the diagnostic criteria
* Patients with β-hCG levels <5000 mIU/ml,
* Patients without serious or persistent abdominal pain
* Patients without fetal cardiac activity observed
* Ectopic mass size smaller than 3-4 cm
* Patients without contraindications for methotrexate and letrozole

Exclusion Criteria:

* Ruptured ectopic pregnancies
* Hemodynamically unstable patients
* Patients with acute abdomen or intra-abdominal bleeding
* Patients with fetal cardiac activity
* β-hCG levels below 500 mIU/mL or above 5000 mIU/mL
* Patients non-compliant with treatment
* Ectopic pregnancy size over 40 mm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Ectopic pregnancy patients are included.
Enrollment: 60 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Decrease in β-hCG levels | On day 1, 4 and 7
  Serum β-hCG titration was monitored on days 1, 4, and 7 using the same laboratory kit.

SECONDARY OUTCOMES:
Need of surgical interventions | On the days of admission.
Hospitalization Days | Through study completion, an average of 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will be shared directly upon reasonable request.